CLINICAL TRIAL: NCT02067468
Title: Evaluation of Strategies for Optimal Clinical Management of Women With Atypical Squamous Cells of Undetermined Significance (ASC-US)
Brief Title: Optimal Strategy for the Management of ASCUS Cytology in Health Care Services of Medellin, Colombia
Acronym: ASCUS-COL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: International Agency for Research on Cancer (Other); Barts and the London School of Medicine and Dentistry (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); QIAGEN Gaithersburg, Inc (Industry); EPS SURA (Unknown); EPS COMFAMA (Unknown); EPS COMFENALCO (Unknown); DINAMICA IPS (Unknown); Laboratorio Clínico Escuela de Microbiología (Universidad de Antioquia) (Unknown); Metrosalud (Unknown)
Responsible Party: Principal Investigator, Gloria I. Sanchez, MSc, PhD, Associate Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 111545921657
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cervical Abnormalities; Cervical Intraepithelial Neoplasia Grade 2/3; Cervical Cancer
Keywords: Human Papillomavirus; cervical cancer; health services research; Colombia; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Human Papillomavirus DNA Tests; Colposcopy; Cytological Techniques; Papanicolaou Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HPV test (Experimental): Women with ASC-US cytology are HPV tested and those HPV positive are refer to Colposcopy
  Interventions: Device: HPV test; Procedure: COLPOSCOPY
- COLPOSCOPY (Active Comparator): Women with ASC-US cytology are immediately refer to colposcopy
  Interventions: Procedure: COLPOSCOPY
- CYTOLOGY (Active Comparator): Women with ASC-US Cytology are follow-up with cytology at 6 and/or 12 months and be referred to colposcopy if any of these cytologies is ASC-US or higher
  Interventions: Procedure: COLPOSCOPY; Device: cytology

INTERVENTIONS:
Device: HPV test — QIAGEN - The Digene HPV test®
  Other Names: Human Papillomavirus test; DNA HPV test; High risk HPV test
  Arms: HPV test
Procedure: COLPOSCOPY — Colposcopy routine health services
Device: cytology — Cytology routine health services
  Other Names: Pap smear; Papanicolaou test; cervical cytology
  Arms: CYTOLOGY

SUMMARY:
Cervical cancer as well cervical preneoplastic abnormalities (CIN2+) are cause by human papillomavirus (HPV) infection. These abnormalities have been historically detected by cervical cytology, but recent evidence shows that HPV testing is superior to cytology to detect cervical lesions that eventually will progress to cancer. Despite evidence, conventional cytology (Pap) remains as a primary screening test in Colombia and HPV test is recommended as a triage test for women with atypical squamous cells of undetermined significance (ASC-US) in settings around the world. Women with ASC-US have low risk to CIN2+ but higher than healthy population, and therefore it is important to provide appropriate clinical management. However, there is no consensus of how to deal women with ASC-US and therefore there are still three strategies for this purpose: 1) immediate colposcopy, 2) repeat conventional cytology at 6 and 12 months and 3) HPV testing. The main objective of this study is to compare the effectiveness and the efficient among the strategies as well as to evaluate the acceptability of the HPV testing in a real-life setting.

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness and efficiency of immediate colposcopy (IC), repeat conventional cytology at 6 and 12 months (RC) and HPV triage (HPV) (QIAGEN-The digene HPV Test®) for the clinical management of women with ASC-US insured in healthcare management organizations (HMO) within the Colombian health security system. This study randomized 2,661 20-69 years old women with ASC-US, insured in HMOs in Medellin-Colombia to 3 arms: IC, RC and HPV. All women are scheduled for a visit at 2 years after recruitment that includes HPV-test/cytology and colposcopy either if HPV+ (RLU>=1) or abnormal cytology (>=ASC-US). This colposcopy is performed by a trained colposcopist and women are followed-up according to a well-defined algorithm. The fewer high-grade cervical neoplasia (CIN2+) rate at the end of following will determine the most effective arm. The most efficiency arm will be which reach the major effective with the minimum resource (cytologies, colposcopies and histologies) consumed. The resource consumed is being retrieved from the HMOs. This study also pretends to evaluate the acceptability of the HPV testing. This study will allow us to know if within the Colombian health security system, the HPV test will remain superior to repeating cytology and/or to immediate colposcopy as it has been demonstrated in randomized controlled trials carried out in outside settings.

ELIGIBILITY:
Inclusion Criteria:

* ASC-US cytology, living in metropolitan area of Medellin

Exclusion Criteria:

* Previous abnormal cytology

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2661 (Actual)
Dates: Start 2011-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria I Sanchez, MSc, PhD, Principal Investigator — Universidad de Antioquia; Armando Baena, MSc, PhD, Study Chair — Universidad de Antioquia; Maria C Agudelo, MD, Study Chair — Universidad de Antioquia; Alejandra Botero, MSc, Study Chair — Universidad de Antioquia; Victor Florez, MSc, Study Chair — Universidad de Antioquia; Calatina Villa, BSc, Study Chair — Universidad de Antioquia; Astrid Bedoya, MSc, Study Chair — Universidad de Antioquia; Guadalupe Posada, MD, Esp, Study Chair — DINAMICA IPS; Carlos A Buitrago, MD, Esp, Study Chair — EPS COMFENALCO; Juan C Ochoa, MD, Esp, Study Chair — EPS COMFAMA; Luis J Gomez, MD, Esp, Study Chair — DINAMICA IPS; Tatiana Ramirez, BSc, Study Chair — Universidad de Antioquia; Maribel Almonte, MSc, PhD, Study Chair — International Agency for Research on Cancer (IARC); Rolando Herrero, MSc, PhD, Study Chair — International Agency for Research on Cancer (IARC); Peter Sasieni, MSc, PhD, Study Chair — Centre for Cancer Prevention, Queen Mary University of London; Yessid Álvarez, Student, Study Chair — Universidad de Antioquia
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] ASCUS-LSIL Traige Study (ALTS) Group. Results of a randomized trial on the management of cytology interpretations of atypical squamous cells of undetermined significance. Am J Obstet Gynecol. 2003 Jun;188(6):1383-92. doi: 10.1067/mob.2003.457. PMID 12824967
- [Background] Andres-Gamboa O, Chicaiza L, Garcia-Molina M, Diaz J, Gonzalez M, Murillo R, Ballesteros M, Sanchez R. Cost-effectiveness of conventional cytology and HPV DNA testing for cervical cancer screening in Colombia. Salud Publica Mex. 2008 Jul-Aug;50(4):276-85. doi: 10.1590/s0036-36342008000400005. PMID 18670718
- [Background] Schiffman M, Adrianza ME. ASCUS-LSIL Triage Study. Design, methods and characteristics of trial participants. Acta Cytol. 2000 Sep-Oct;44(5):726-42. doi: 10.1159/000328554. PMID 11015972
- [Background] Schiffman M, Solomon D. Findings to date from the ASCUS-LSIL Triage Study (ALTS). Arch Pathol Lab Med. 2003 Aug;127(8):946-9. doi: 10.5858/2003-127-946-FTDFTA. PMID 12873166
- [Background] Arbyn M, Sasieni P, Meijer CJ, Clavel C, Koliopoulos G, Dillner J. Chapter 9: Clinical applications of HPV testing: a summary of meta-analyses. Vaccine. 2006 Aug 31;24 Suppl 3:S3/78-89. doi: 10.1016/j.vaccine.2006.05.117. PMID 16950021
- [Background] Carozzi FM, Confortini M, Cecchini S, Bisanzi S, Cariaggi MP, Pontenani G, Raspollini MR, Sani C, Zappa M, Ciatto S. Triage with human papillomavirus testing of women with cytologic abnormalities prompting referral for colposcopy assessment. Cancer. 2005 Feb 25;105(1):2-7. doi: 10.1002/cncr.20736. PMID 15593261
- [Background] Legood R, Gray A, Wolstenholme J, Moss S. Lifetime effects, costs, and cost effectiveness of testing for human papillomavirus to manage low grade cytological abnormalities: results of the NHS pilot studies. BMJ. 2006 Jan 14;332(7533):79-85. doi: 10.1136/bmj.38698.458866.7C. Epub 2006 Jan 6. PMID 16399769
- [Background] Kulasingam SL, Kim JJ, Lawrence WF, Mandelblatt JS, Myers ER, Schiffman M, Solomon D, Goldie SJ; ALTS Group. Cost-effectiveness analysis based on the atypical squamous cells of undetermined significance/low-grade squamous intraepithelial lesion Triage Study (ALTS). J Natl Cancer Inst. 2006 Jan 18;98(2):92-100. doi: 10.1093/jnci/djj009. PMID 16418511
- [Background] Sheriff SK, Petry KU, Ikenberg H, Crouse G, Mazonson PD, Santas CC. An economic analysis of human papillomavirus triage for the management of women with atypical and abnormal Pap smear results in Germany. Eur J Health Econ. 2007 Jun;8(2):153-60. doi: 10.1007/s10198-007-0038-5. Epub 2007 Feb 17. PMID 17308921
- [Background] Vanni T, Legood R, Franco EL, Villa LL, Luz PM, Schwartsmann G. Economic evaluation of strategies for managing women with equivocal cytological results in Brazil. Int J Cancer. 2011 Aug 1;129(3):671-9. doi: 10.1002/ijc.25708. Epub 2010 Nov 12. PMID 20886598
- [Background] Dillner L, Kemetli L, Elfgren K, Bogdanovic G, Andersson P, Carlsten-Thor A, Andersson S, Persson E, Rylander E, Grillner L, Dillner J, Tornberg S. Randomized healthservices study of human papillomavirus-based management of low-grade cytological abnormalities. Int J Cancer. 2011 Jul 1;129(1):151-9. doi: 10.1002/ijc.25649. Epub 2010 Nov 9. PMID 20824706
- [Background] Ostensson E, Froberg M, Hjerpe A, Zethraeus N, Andersson S. Economic analysis of human papillomavirus triage, repeat cytology, and immediate colposcopy in management of women with minor cytological abnormalities in Sweden. Acta Obstet Gynecol Scand. 2010 Oct;89(10):1316-25. doi: 10.3109/00016349.2010.512066. PMID 20846064
- [Background] Inter-American-Development-Bank. Structured Pluralism: Toward an Innovative Model for the Reform of Health Systems in Latin America. Office of the Chief Economist. 1997;Working Paper 353.
- [Background] Luce BR, Kramer JM, Goodman SN, Connor JT, Tunis S, Whicher D, Schwartz JS. Rethinking randomized clinical trials for comparative effectiveness research: the need for transformational change. Ann Intern Med. 2009 Aug 4;151(3):206-9. doi: 10.7326/0003-4819-151-3-200908040-00126. Epub 2009 Jun 30. No abstract available. PMID 19567619
- [Background] Verdoodt F, Szarewski A, Halfon P, Cuschieri K, Arbyn M. Triage of women with minor abnormal cervical cytology: meta-analysis of the accuracy of an assay targeting messenger ribonucleic acid of 5 high-risk human papillomavirus types. Cancer Cytopathol. 2013 Dec;121(12):675-87. doi: 10.1002/cncy.21325. Epub 2013 Jul 23. PMID 23881840
- [Background] Arbyn M, Ronco G, Anttila A, Meijer CJ, Poljak M, Ogilvie G, Koliopoulos G, Naucler P, Sankaranarayanan R, Peto J. Evidence regarding human papillomavirus testing in secondary prevention of cervical cancer. Vaccine. 2012 Nov 20;30 Suppl 5:F88-99. doi: 10.1016/j.vaccine.2012.06.095. PMID 23199969
- [Background] Sorbye SW, Arbyn M, Fismen S, Gutteberg TJ, Mortensen ES. Triage of women with low-grade cervical lesions--HPV mRNA testing versus repeat cytology. PLoS One. 2011;6(8):e24083. doi: 10.1371/journal.pone.0024083. Epub 2011 Aug 30. PMID 21918682
- [Background] Arbyn M, Martin-Hirsch P, Buntinx F, Van Ranst M, Paraskevaidis E, Dillner J. Triage of women with equivocal or low-grade cervical cytology results: a meta-analysis of the HPV test positivity rate. J Cell Mol Med. 2009 Apr;13(4):648-59. doi: 10.1111/j.1582-4934.2008.00631.x. Epub 2009 Jan 23. PMID 19166485
- [Background] Cuzick J, Arbyn M, Sankaranarayanan R, Tsu V, Ronco G, Mayrand MH, Dillner J, Meijer CJ. Overview of human papillomavirus-based and other novel options for cervical cancer screening in developed and developing countries. Vaccine. 2008 Aug 19;26 Suppl 10:K29-41. doi: 10.1016/j.vaccine.2008.06.019. PMID 18847555
- [Background] Dalla Palma P, Pojer A, Girlando S. HPV triage of women with atypical squamous cells of undetermined significance: a 3-year experience in an Italian organized programme. Cytopathology. 2005 Feb;16(1):22-6. doi: 10.1111/j.1365-2303.2004.00196.x. PMID 15859311
- [Background] Instituto Nacional de C. Recomendaciones para el tratamiento de las pacientes con citologia reportada con células escamosas atipicas de significado indeterminado (ASC-US) en Colombia. Guias de practica clinica (No. 2). Bogota, Colombia: INC, 2007
- [Result] Baena A, Agudelo MC, Posada G, Lopez C, Buitrago CA, Suescun D, Gomez LJ, Ochoa JC, Sasieni P, Almonte M, Herrero R, Sanchez GI. Efectividad de tres estrategias para el manejo clínico de la citología ASC-US en servicios rutinarios de salud de Medellín, Colombia: diseño y resultados de dos años de seguimiento del ensayo pragmático aleatorio ASCUS-COL (NCT02067468). Rev Colomb Cancerol 2017;21:49 - DOI: 10.1016/j.rccan.2017.02.012
- [Result] Baena A, Agudelo MC, Posada G, Lopez C, Buitrago CA, Suescun D, Gomez LJ, Ochoa JC, Sasieni P, Almonte M, Herrero R, Sanchez GI. EI triage con prueba de VPH de aIto riesgo y Ia citoIogía repetida son estrategias eficientes para eI manejo cIínico de mujeres con citoIogía ASC-US en servicios rutinarios de saIud de MedeIIín, CoIombia: resuItados finaIes deI ensayo pragmático aIeatorio ASCUS-COL. Rev Colomb Cancerol 2017;21:49-50 - DOI: 10.1016/j.rccan.2017.02.013
- [Derived] Urrea Cosme Y, Cordoba Sanchez V, Sanchez GI, Baena A, Ruiz Osorio MA, Rodriguez Zabala D, Garces-Palacio IC. Health-related quality of life of women after HPV testing as triage strategy for an abnormal Pap smear: a nested randomized pragmatic trial in a middle-income country. Qual Life Res. 2020 Nov;29(11):2999-3008. doi: 10.1007/s11136-020-02563-w. Epub 2020 Jul 2. PMID 32617889
- [Derived] Henao AR, Gomez NEM, Gonzalez-Gomez D, Garces-Palacio IC. Validation of Spanish version of the human papilloma virus impact profile (HIP). Curr Med Res Opin. 2020 Apr;36(4):705-712. doi: 10.1080/03007995.2020.1729709. Epub 2020 Mar 6. PMID 32049551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After a great effort, due to logistic issues, it was only possible to enroll 2661 participants instead of 3000 as it had been stated in the submitted protocol. Despite it, the trial had enough statistical power to answer the research questions.
Groups:
- COLPOSCOPY: Women with ASC-US cytology are immediately referred to colposcopy
  COLPOSCOPY: Colposcopy routine health services
Period: Overall Study
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Started | 882 | 890 | 889
Followed-up Through Medical Records (All included women followed through databases and medical records manually ascertained from HMOs) | 882 | 890 | 889
Had at Least One Routine Colposcopy (Referred to colposcopy: 100% for COLPOSCOPY, abnormal Pap for CYTOLOGY (31%), and HPV+ for HPV (41%)) | 772 | 372 | 462
Completed | 882 | 890 | 889
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HPV Test: Women with ASC-US cytology are HPV tested and those HPV positive are referred to Colposcopy
  HPV test: QIAGEN - The Digene HPV test®
  COLPOSCOPY: Colposcopy routine health services
- Total: Total of all reporting groups
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test | Total
Number analyzed (Participants) | 882 | 890 | 889 | 2661
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (11) | 37 (11) | 37.4 (10.9) | 37.3 (11)
Age, Customized [Count of Participants; unit: Participants]
  Age, years: 20-30 | 290 | 305 | 289 | 884
  Age, years: 31-40 | 240 | 248 | 233 | 721
  Age, years: 41-50 | 239 | 225 | 261 | 725
  Age, years: 51-69 | 113 | 112 | 106 | 331
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 882 | 890 | 889 | 2661
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 882 | 890 | 889 | 2661
Healthcare Management Organization (Secondary centers) [Count of Participants; unit: Participants] — This measure refers to the number of participants enrolled from three different Healthcare Management Organizations (HMOs) of the two national health insurance schemes (two from the contributory health regime and one from the subsidized regime). To guarantee the anonymity of HMOs, these were labeled as HMO #1, HMO #2, and HMO #3. In total, 636 women were included from HMO #1, 1364 from HMO #2, and 661 from HMO #3.
  Participants
    Healthcare Management Organization #1 | 196 | 233 | 207 | 636
    Healthcare Management Organization #2 | 461 | 442 | 461 | 1364
    Healthcare Management Organization #3 | 225 | 215 | 221 | 661
Marital Satus [Count of Participants; unit: Participants]
  Married/cohabiting | 420 | 440 | 446 | 1306
  Divorced/separated | 70 | 83 | 83 | 236
  Widowed | 31 | 34 | 25 | 90
  Single | 361 | 333 | 335 | 1029
Education [Count of Participants; unit: Participants]
  Complete/some elementary school | 220 | 236 | 246 | 702
  Complete/some secondary school | 426 | 430 | 418 | 1274
  Technician | 150 | 147 | 144 | 441
  Professional or higher | 86 | 77 | 81 | 244
Frequency of cytology use [Count of Participants; unit: Participants]
  Once or more than once every year | 608 | 593 | 590 | 1791
  Once every 2-3 years | 174 | 181 | 176 | 531
  Once every 4-5 years | 54 | 59 | 64 | 177
  Once every 6-10 years | 24 | 25 | 22 | 71
  Less than once every 10 years | 6 | 6 | 9 | 21
  Do not know/Do not answer | 16 | 26 | 28 | 70

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Participants Diagnosed by the Community Pathologist With Cervical Intraepithelial Neoplasia Grade 2 or Higher (CIN2+): "Community-based CIN2+"
Description: Cumulative Cervical Intraepithelial Neoplasia Grade 2 or higher (CIN2+) diagnosed by the community pathologists during the two years of follow-up. The first community-based CIN2+ diagnosis was adjudicated to the participant (including the exit visit if none community-based CIN2+ during the two years of follow-up). This outcome is used for the effectiveness analysis of the three strategies.
Time Frame: Two years since the enrolment to the exit visit (inclusive)
Population: Cumulative cases of CIN2+ diagnosed by the community pathologists from the healthcare institutions according to arm
Measure: Count of Participants; unit: Participants
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 882 | 890 | 889
Participants
  Community-based <CIN2 | 847 | 835 | 848
  Community-based CIN2 | 30 | 43 | 31
  Community-based CIN3 | 4 | 11 | 10
  Community-based Cancer | 1 | 1 | 0

2. Secondary Outcome: Cumulative Number of Participants Diagnosed by a Panel of External Experts With Cervical Intraepithelial Neoplasia Grade 2 or Higher (CIN2+): "Reviewed CIN2+"
Description: Cumulative Cervical Intraepithelial Neoplasia Grade 2 or higher (CIN2+) diagnosed by a panel of external experts obtained after histological review of biopsies emitted by the community pathologists. Biopsies obtained during the two years of follow-up and the exit visit were reviewed by a panel of two external experts and a final result was adjudicated to each participant based on the panel of experts and the community of pathologists. This outcome is used for the effectiveness analysis of the three strategies.
Time Frame: Two years since the enrolment to the exit visit (inclusive)
Population: Cumulative cases of CIN2+ diagnosed by a panel of external expert pathologists according to arm
Measure: Count of Participants; unit: Participants
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 882 | 890 | 889
Participants
  Reviewed <CIN2 | 813 | 809 | 827
  Reviewed CIN2 | 51 | 61 | 48
  Reviewed CIN3 | 16 | 18 | 14
  Reviewed Cancer | 2 | 2 | 0

3. Secondary Outcome: Number of Participants Diagnosed by a Panel of External Experts With Cervical Intraepithelial Neoplasia Grade 2 or Higher (CIN2+) at the Exit Visit, Two Years After the Enrolment: "Exit-reviewed CIN2+"
Description: Cervical Intraepithelial Neoplasia Grade 2 or higher (CIN2+) diagnosed by a panel of external experts after reviewing biopsies collected at the exit visit, two years after the enrolment. This outcome is an estimate of the remaining disease that was not detected by the strategies during the 2 years of follow-up. The outcome was obtained after the review of all the biopsies taken during the exit visit. Biopsies were taken using a standardized research protocol to ensure the completeness of the remaining disease. Basically, all women attending the exit visit were tested with HPV testing and Pap and referred to colposcopy if any HPV positive or abnormal cytology. The colposcopy was performed by a researcher of the study team who took up to two biopsies from the observed lesion plus one or two at random if none lesion was observed. All biopsies were reviewed by the external panel. This outcome is used for the efficiency analysis of the three strategies.
Time Frame: Exit visit (two years after the enrolment)
Population: Exit-reviewed CIN2+ detected at the exit visit (2 years after the enrolment) of women with ASC-US cytology stratified by arm
Measure: Count of Participants; unit: Participants
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 882 | 890 | 889
Participants
  Exit-reviewed <CIN2 | 852 | 851 | 866
  Exit-reviewed CIN2+ | 30 | 39 | 23

4. Secondary Outcome: Number of Clinical Records (Cytologies, Colposcopies, and Histologies): "Health Care Utilization"
Description: The outcome is defined as the number of cytologies, colposcopies, and histologies routinely performed during the two years of follow-up. Records were identified in databases or manually searched from clinical records. This outcome will be used for the analysis of the efficiency of the three strategies.
Time Frame: Two years since the enrolment to before the exit visit (i.e., excluding clinical records collected at the exit visit)
Population: Utilization of cytology, colposcopy and histology during the routine follow-up of women with ASC-US cytology stratified by arm
Measure: Number; unit: Clinical records
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 882 | 890 | 889
Clinical records
  Cytology utilization | 904 | 1218 | 816
  Colposcopy utilization | 964 | 509 | 633
  Histology utilization | 572 | 349 | 401
  Total utilization | 2440 | 2076 | 1850

5. Secondary Outcome: Self-esteem
Description: Self-esteem corresponds to the self-assessment of a positive or negative evaluation toward oneself. This outcome was measured using the Rosenberg Scale through 10 Likert-type questions with scores varying between 1 and 4 (1=strongly agree, 2=agree, 3=disagree, 4=strongly disagree). Total values range between 10 and 40 where lower scores suggest lower self-esteem. This outcome was measured at the enrollment visit, between two weeks and two months after receiving the triage result, and after one year of receiving the triage result.
Time Frame: Two years between the enrolment and the exit visit
Population: This is a nested analysis that included 394 subjects of the ASCUS-COL trial (142 in COLPOSCOPY, 103 in CYTOLOGY, and 149 HPV) who accepted to participate and completed the follow-up of three measurements over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 142 | 103 | 149
score on a scale
  Self-esteem at enrollment | 32.9 (4.40) | 33.0 (4.25) | 32.8 (4.17)
  Self-esteem after receiving the triage result | 34.8 (4.84) | 33.9 (4.38) | 34.4 (4.78)
  Self-esteem after one year of the triage result | 35.4 (4.43) | 35.5 (5.26) | 35.2 (4.84)

6. Secondary Outcome: Trait Anxiety
Description: Trait anxiety refers to the sustainable tendency to experience negative emotions (such as fears, worries, and anxiety) in various situations. This outcome was measured using the Spielberger State-Trait-Anxiety Inventory (STAI) through 20 Likert-type questions with scores varying between 0 and 3 (0=not at all, 1=somewhat, 2=moderately, 3=very much). Total values range between 0 and 60 where higher scores suggest higher levels of anxiety. This outcome was measured at the enrollment visit, between two weeks and two months after receiving the triage result, and after one year of receiving the triage result.
Time Frame: Two years between the enrolment and the exit visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 142 | 103 | 149
score on a scale
  Trait anxiety at enrollment | 17.5 (13.27) | 17.4 (11.34) | 17.7 (11.10)
  Trait anxiety after receiving the triage result | 16.3 (13.14) | 16.8 (12.08) | 17.7 (12.80)
  Trait anxiety after one year of the triage result | 14.9 (11.95) | 13.4 (11.15) | 14.9 (12.51)

7. Secondary Outcome: State Anxiety
Description: State anxiety refers to the transitory tendency to experience negative emotions (such as fears, worries, and anxiety). This outcome was measured using the Spielberger State-Trait-Anxiety Inventory (STAI) through 20 Likert-type questions with scores varying between 0 and 3 (0=not at all, 1=somewhat, 2=moderately, 3=very much). Total values range between 0 and 60 where higher scores suggest higher levels of anxiety. This outcome was measured at the enrollment visit, between two weeks and two months after receiving the triage result, and after one year of receiving the triage result.
Time Frame: Two years between the enrolment and the exit visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 142 | 103 | 149
score on a scale
  State anxiety at enrollment | 15.3 (13.23) | 13.6 (11.03) | 14.3 (11.45)
  State anxiety after receiving the triage result | 14.1 (14.11) | 13.4 (12.55) | 14.1 (13.65)
  State anxiety after one year of the triage result | 9.8 (10.79) | 10.8 (11.76) | 9.5 (11.38)

8. Secondary Outcome: Concerns About Fertility, Cancer, and Gynecological Health
Description: This outcome was measured using the HPV Impact Profile (HIP) scale through the following five domains: concerns about cancer and loss of fertility; emotional impact (depression and anxiety); self-image; interaction with the medical staff (pain or discomfort during the visit); and impact upon the life and its control. The response to each domain was measured on a scale from 0 to 10 (0=not at all, 1-3=a little, 4-6=somewhat, 7-9=a great deal, 10=extremely) and was then transformed to a scale from 0 to 100. A total score was calculated by adding all the items. Values <40 indicate no or little impact, between 40 and 70 moderate impact, and >70 indicate high psychosocial impact. This outcome was measured at the enrollment visit, between two weeks and two months after receiving the triage result, and after one year of receiving the triage result.
Time Frame: Two years between the enrolment and the exit visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
Number analyzed (Participants) | 142 | 103 | 149
score on a scale
  Concerns at enrollment | 35.3 (15.23) | 38.1 (15.45) | 36.0 (14.72)
  Concerns after receiving the triage result | 25.0 (16.48) | 25.7 (15.42) | 27.2 (18.11)
  Concerns after one year of the triage result | 18.7 (13.07) | 18.4 (14.38) | 17.9 (12.79)

ADVERSE EVENTS:
Time Frame: Since the enrolment to the exit visit (2 years after the enrolment)
Arm/Group | COLPOSCOPY | CYTOLOGY | HPV Test
All-Cause Mortality (participants affected / at risk) | 0/882 | 0/890 | 0/889
Serious Adverse Events (participants affected / at risk) | 0/882 | 0/890 | 0/889
Other Adverse Events (participants affected / at risk) | 0/882 | 0/890 | 0/889

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No